CLINICAL TRIAL: NCT04352634
Title: The Impact of the Covid-19 Pandemic on the Mental Health of Workers in Health Services: The Covid-19 HEalth caRe wOrkErS (HEROES) Study
Brief Title: The Covid-19 HEalth caRe wOrkErS (HEROES) Study
Acronym: HEROES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Rubén Alvarado, PhD, University of Chile
Other Study IDs: HEROES Covid-19
Record Dates: First submitted 2020-04-08; First posted 2020-04-20 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid-19; Mental Health Disorder; Stress Disorder; Anxiety; Depression; SARS-CoV-2
Keywords: Covid-19; healthcare professionals; mental health; pandemic
MeSH Terms: conditions — COVID-19; Mental Disorders; Stress Disorders, Traumatic; Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Workers who interact with people with confirmed or suspected COVID-19 at different health services (primary care centers, emergency units, specialized care units, inpatient care units, critically ill patient units, among others). Potential participants will include any type of worker in these centers, including clinical and administrative staff, as well as supportive staff (e.g., food services)
  Interventions: Other: Exposure to the SARS-CoV-2 and its consequences

INTERVENTIONS:
Other: Exposure to the SARS-CoV-2 and its consequences — This is an observational design. Participants are exposed to the SARS-CoV-2, the Covid-19 pandemic, and/or its consequences

SUMMARY:
Since December 2019 the world has been shaken with an enormous global threat: the Covid-19 pandemic. This new kind of coronavirus is generating an unprecedented impact both on the general population and on the healthcare systems in most countries. Health services are trying to expand their capacity to respond to the pandemic, taking actions such as increasing the number of beds; acquiring necessary equipment to provide intensive therapy (ventilators), and calling retired health professionals and health students so they can assist the overwhelmed health care workforce. Unfortunately, these organizational changes at health facilities, along with the fears and concerns of becoming ill with the virus or infecting their families, put an enormous emotional burden on workers in health services which may lead to negative outcomes on mental health in this population.

Recent cross-sectional studies in China indicate that health service workers exposed to people with Covid-19 reported higher rates of depressive and anxious symptoms. This negative impact on mental health among health workers in China has also been informally reported in other countries where the Covid-19 pandemic has been devastating in its effects (such as Spain and Italy), as well as in countries where the pandemic is becoming a growing public health problem. This is particularly relevant in regions with fewer resources (Latin America, North Africa), where there are limited means and the response from the health system is usually insufficient. Moreover, it is necessary to study these negative effects longitudinally considering that some effects will appear over time (post-traumatic stress).

The COVID-19 HEalth caRe wOrkErS (HEROES) study is a large, bottom-up, South-North initiative aimed to evaluate the impact of the COVID-19 pandemic on the mental health of health care workers (HCWs). HEROES encompasses a wide variety of academic institutions in 19 LMICs and 8 HICs, in partnership with the Pan American Health Organization (PAHO) and with support from the World Health Organization (WHO). The HEROES study is led by Dr. Rubén Alvarado at University of Chile, and Dr. Ezra Susser and Franco Mascayano at Columbia U Mailman School of Public Health.

DETAILED DESCRIPTION:
Since December 2019 the world has been shaken with an enormous global threat: the Covid-19 pandemic. This new kind of coronavirus is generating an unprecedented impact both on the general population and on the healthcare systems in most countries. Health services are trying to expand their capacity to respond to the pandemic, taking actions such as increasing the number of beds; acquiring necessary equipment to provide intensive therapy (ventilators), and calling retired health professionals and health students so they can assist the overwhelmed health care workforce. Unfortunately, these organizational changes at health facilities, along with the fears and concerns of becoming ill with the virus or infecting their families, put an enormous emotional burden on workers in health services which may lead to negative outcomes on mental health in this population. Based on the literature to date, Covid-19 is significantly larger than previous pandemics in terms of the number of affected people worldwide, its spread across countries, its impact on healthcare systems and the severity of measures that have been taken by governments. Immediate consequences are palpable in the health care system. Many healthcare workers are overwhelmed by the increased workload; the lack of supplies and materials to provide appropriate treatment; the lack of clinical guidelines on prioritization and triage; and the increased feelings of isolation and loneliness. Previous research indicates that these negative effects can last over time and lead to the development of serious mental health problems such as post-traumatic stress disorder.

Recent cross-sectional studies in China indicate that health service workers exposed to people with Covid-19 reported higher rates of depressive and anxious symptoms. This negative impact on mental health among health workers in China has also been informally reported in other countries where the Covid-19 pandemic has been devastating in its effects (such as Spain and Italy), as well as in countries where the pandemic is becoming a growing public health problem. This is particularly relevant in regions with fewer resources (Latin America, North Africa), where there are limited means and the response from the health system is usually insufficient. Moreover, it is necessary to study these negative effects longitudinally considering that some effects will appear over time (post-traumatic stress). Also, it is necessary to take into account the nature and the extent of the health response (e.g., deployment, increased workload) in order to advance our understanding of these complex phenomenon and to inform policy and develop the kind of supports that this population deems useful.

The COVID-19 HEalth caRe wOrkErS (HEROES) study is a large, bottom-up, South-North initiative aimed to evaluate the impact of the COVID-19 pandemic on the mental health of health care workers (HCWs). HEROES encompasses a wide variety of academic institutions in 19 LMICs and 8 HICs, in partnership with the Pan American Health Organization (PAHO) and with support from the World Health Organization (WHO). The HEROES study is led by Dr. Rubén Alvarado at University of Chile, and Dr. Ezra Susser and Franco Mascayano at Columbia U Mailman School of Public Health.

Participants will complete an online questionnaire, which will be completely self-administered. It will take approximately 12 minutes and includes sociodemographic data, questions on work activity, training, fears and concerns related to Covid-19, as well as the GHQ-12 and a series of questions on other mental health issues (e.g., suicide, acute stress), resilience and psycho/social factors (e.g., formal and informal support).

ELIGIBILITY:
Inclusion Criteria:

* Legal age
* Currently working on a health service that provides care to COVID-19 patients
* Give informed consent

Exclusion Criteria:

* Inability to use electronic devices (required to complete the survey)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include workers who interact with people with confirmed or suspected COVID-19 at different health services (primary care centers, emergency units, specialized care units, inpatient care units, critically ill patient units, among others). Potential participants will include any type of worker in these centers, including clinical and administrative staff, as well as supportive staff (e.g., food services)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-26 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depressive symptoms | 12 months
  The 12-item version of the General Health Questionnaire (GHQ-12) is a self-reported instrument that measures symptoms of anxiety and depression. It provides cut-off points to identify people at risk of anxiety and/or depression, which differ slightly between countries

SECONDARY OUTCOMES:
Experiences, fears and concerns about the Covid-19 | Baseline
  Ad hoc survey on experiences, fears, and concerns about Covid-19
Experiences, fears and concerns about the Covid-19 | 3 months
  Ad hoc survey on experiences, fears, and concerns about Covid-19
Experiences, fears and concerns about the Covid-19 | 6 months
  Ad hoc survey on experiences, fears, and concerns about Covid-19
Experiences, fears and concerns about the Covid-19 | 12 months
  Ad hoc survey on experiences, fears, and concerns about Covid-19
Training and resource prioritization | Baseline
  Ad hoc survey on Covid-19 training and resource prioritization
Training and resource prioritization | 3 months
  Ad hoc survey on Covid-19 training and resource prioritization
Training and resource prioritization | 6 months
  Ad hoc survey on Covid-19 training and resource prioritization
Training and resource prioritization | 12 months
  Ad hoc survey on Covid-19 training and resource prioritization
Suicide ideation (presence) | Baseline
  Item from the Columbia Suicide Severity Rating Scale (C-SSRS) that measures suicidal ideation with a dichotomous answer (presence/absence)
Suicide ideation (presence) | 3 months
  Item from the Columbia Suicide Severity Rating Scale (C-SSRS) that measures suicidal ideation with a dichotomous answer (presence/absence)
Suicide ideation (presence) | 6 months
  Item from the Columbia Suicide Severity Rating Scale (C-SSRS) that measures suicidal ideation with a dichotomous answer (presence/absence)
Suicide ideation (presence) | 12 months
  Item from the Columbia Suicide Severity Rating Scale (C-SSRS) that measures suicidal ideation with a dichotomous answer (presence/absence)
Suicide ideation (frequency) | Baseline
  5-point Likert item from the Columbia Suicide Severity Rating Scale (C-SSRS). Higher scores indicate higher frequency.
Suicide ideation (frequency) | 3 months
  5-point Likert item from the Columbia Suicide Severity Rating Scale (C-SSRS). Higher scores indicate higher frequency.
Suicide ideation (frequency) | 6 months
  5-point Likert item from the Columbia Suicide Severity Rating Scale (C-SSRS). Higher scores indicate higher frequency.
Suicide ideation (frequency) | 12 months
  5-point Likert item from the Columbia Suicide Severity Rating Scale (C-SSRS). Higher scores indicate higher frequency.
Acute stress symptoms | Baseline
  Ad hoc 3-item survey to evaluate acute stress disorder. Higher values of the 5-points Likert scales suggest higher frequency of symptoms
Acute stress symptoms | 3 months
  Ad hoc 3-item survey to evaluate acute stress disorder. Higher values of the 5-points Likert scales suggest higher frequency of symptoms
Acute stress symptoms | 6 months
  Ad hoc 3-item survey to evaluate acute stress disorder. Higher values of the 5-points Likert scales suggest higher frequency of symptoms
Acute stress symptoms | 12 months
  Ad hoc 3-item survey to evaluate acute stress disorder. Higher values of the 5-points Likert scales suggest higher frequency of symptoms
Psycho/social support and network | Baseline
  Ad hoc survey on support network. The answers to the multiple items will be adjusted so higher values indicate higher levels of psychological and social support
Psycho/social support and network | 3 months
  Ad hoc survey on support network. The answers to the multiple items will be adjusted so higher values indicate higher levels of psychological and social support
Psycho/social support and network | 6 months
  Ad hoc survey on support network. The answers to the multiple items will be adjusted so higher values indicate higher levels of psychological and social support
Psycho/social support and network | 12 months
  Ad hoc survey on support network. The answers to the multiple items will be adjusted so higher values indicate higher levels of psychological and social support
Resilience | Baseline
  The Brief Resilience Scale (BRS) is a 6-item self-reported instrument that measures resilience. The range of scores is 6-30. Higher scores indicate higher resilience levels.
Resilience | 3 months
  The Brief Resilience Scale (BRS) is a 6-item self-reported instrument that measures resilience. The range of scores is 6-30. Higher scores indicate higher resilience levels.
Resilience | 6 months
  The Brief Resilience Scale (BRS) is a 6-item self-reported instrument that measures resilience. The range of scores is 6-30. Higher scores indicate higher resilience levels.
Resilience | 12 months
  The Brief Resilience Scale (BRS) is a 6-item self-reported instrument that measures resilience. The range of scores is 6-30. Higher scores indicate higher resilience levels.
Anxiety and depressive symptoms | Baseline
  The 12-item version of the General Health Questionnaire (GHQ-12) is a self-reported instrument that measures symptoms of anxiety and depression. It provides cut-off points to identify people at risk of anxiety and/or depression, which differ slightly between countries
Anxiety and depressive symptoms | 3 months
  The 12-item version of the General Health Questionnaire (GHQ-12) is a self-reported instrument that measures symptoms of anxiety and depression. It provides cut-off points to identify people at risk of anxiety and/or depression, which differ slightly between countries
Anxiety and depressive symptoms | 6 months
  The 12-item version of the General Health Questionnaire (GHQ-12) is a self-reported instrument that measures symptoms of anxiety and depression. It provides cut-off points to identify people at risk of anxiety and/or depression, which differ slightly between countries

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Alvarado, PhD, Principal Investigator — University of Chile [Universidad de Chile]; Ezra Susser, MD DrPH, Principal Investigator — Columbia University; Franco Mascayano, MPH, Principal Investigator — Columbia Universty
Locations (22):
- Columbia University, New York, New York, United States
- Universidad del Chubut, Rawson, Chubut Province, Argentina
- National Institute of Health Named After Academician S. Avdalbekyan, Yerevan, Armenia
- University of Sydney, Sydney, New South Wales, Australia
- Salud Global, Sucre, Chuquisaca Department, Bolivia
- University of Chile, Santiago, Chile
- Universidad Nacional de Costa Rica, Heredia, Costa Rica
- Society for Emergecy and Disaster Medicine CzMA JEP, Kladno, Bohemia, Czechia
- Hochschule Emden/Leer, Emden, Lower Saxony, Germany
- Centro de Investigaciones de las Ciencias de la Salud -CICS- Facultad de Ciencias Médicas Universidad de San Carlos de Guatemala -USAC-, Guatemala City, Guatemala
- Italy (2):
  - University of Cagliari, Cagliari, CA
  - University of Cagliari, Cagliari
- The Institute for Development Research Advocacy and Applied Care (IDRAAC), Beirut, Lebanon
- Logotipo del comercio Instituto Jalisciense De Salud Mental (SALME), Guadalajara, Jalisco, Mexico
- Maastricht University, Maastricht, Limburg, Netherlands
- University of Ibadan, Ibadan, Oyo State, Nigeria
- Ponce Health Sciences University, Ponce, Puerto Rico
- King Abdullah International medical research center, Riyadh, Central, Saudi Arabia
- Hospital La Paz Institute for Health Research (IdiPAZ), Madrid, Spain
- Razi Hospital La Manouba, Tunis, La Manouba, Tunisia
- Koc University, Istanbul, Sariyer, Turkey (Türkiye)
- PNFA Salud Colectiva Instituto de Altos Estudios Dr Arnoldo Gabaldon, Maracay, Aragua, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] Nacoti M, et al. At the Epicenter of the Covid-19 Pandemic and Humanitarian Crises in Italy: Changing Perspectives on Preparation and Mitigation. NEJM Catalyst, 2020;1(2)
- [Background] Huang L, Lei W, Xu F, Liu H, Yu L. Emotional responses and coping strategies in nurses and nursing students during Covid-19 outbreak: A comparative study. PLoS One. 2020 Aug 7;15(8):e0237303. doi: 10.1371/journal.pone.0237303. eCollection 2020. PMID 32764825
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Derived] Asaoka H, Watanabe K, Miyamoto Y, Restrepo-Henao A, van der Ven E, Moro MF, Alnasser LA, Ayinde O, Balalian AA, Basagoitia A, Durand-Arias S, Eskin M, Fernandez-Jimenez E, Ines FFM, Gimenez L, Hoek HW, Jaldo RE, Lindert J, Maldonado H, Martinez-Ales G, Mediavilla R, McCormack C, Narvaez J, Ouali U, Barrera-Perez A, Calgua-Guerra E, Ramirez J, Rodriguez AM, Seblova D, da Silva ATC, Valeri L, Gureje O, Ballester D, Carta MG, Isahakyan A, Jamoussi A, Seblova J, Solis-Soto MT, Alvarado R, Susser E, Mascayano F, Nishi D; HEROES group. Association of depressive symptoms with incidence and mortality rates of COVID-19 over 2 years among healthcare workers in 20 countries: multi-country serial cross-sectional study. BMC Med. 2024 Sep 12;22(1):386. doi: 10.1186/s12916-024-03585-8. PMID 39267052